CLINICAL TRIAL: NCT01288027
Title: A Phase 4 Prospective Exploratory Muscle Biopsy, Biomarker, and Imaging Assessment Study in Patients With Late-Onset Pompe Disease Treated With Alglucosidase Alfa
Brief Title: Exploratory Muscle Biopsy Assessment Study in Patients With Late-Onset Pompe Disease Treated With Alglucosidase Alfa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU07310; 2010-020611-36 (EudraCT Number); MSC12823 (Other: Sanofi)
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Pompe Disease (Late-Onset); Glycogen Storage Disease Type II (GSD II); Glycogenesis 2 Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alglucosidase Alfa (Experimental)
  Interventions: Biological: Alglucosidase Alfa

INTERVENTIONS:
Biological: Alglucosidase Alfa — Alglucosidase alfa intravenous infusion 20 milligram per kilogram (mg/kg) every other week for 24 weeks.
  Other Names: GZ419829; Myozyme®; Lumizyme®

SUMMARY:
This is an open-label, multicenter study of participants with late-onset Pompe disease naive to treatment with enzyme replacement therapy (ERT). The primary objective of this study is to evaluate glycogen clearance in muscle tissue samples collected pre and post alglucosidase alfa treatment in participants with Late-Onset Pompe disease.

The secondary objectives are to characterize the disease burden in participants with late-onset Pompe disease and explore imaging, histologic, and functional assessments in these participants and to explore potential plasma or urine biomarkers relative to late-onset Pompe disease and participant's response to treatment with alglucosidase alfa (Myozyme®/Lumizyme®/GZ419829).

ELIGIBILITY:
Inclusion Criteria:

* The participant has confirmed acid alpha-glucosidase (GAA) enzyme deficiency from any tissue source and/or confirmed GAA gene mutations and without known cardiac hypertrophy
* The participant is able to ambulate a distance without stopping and without an assistive device. Use of assistive device for community ambulation is appropriate
* The participant has a certain forced vital capacity (FVC) in upright position
* The participant, if female and of childbearing potential, must have a negative pregnancy test (urine beta-human chorionic gonadotropin [beta-hCG]) at baseline

Exclusion Criteria:

* The participant has had previous treatment with ERT
* The participant is wheelchair dependent
* The participant requires invasive-ventilation (non-invasive ventilation is allowed)
* The participant is participating in another clinical study using investigational treatment
* The participant cannot submit to magnetic resonance imaging (MRI) examination because of a formal contraindication such as a pacemaker, implanted ferromagnetic metals, etc
* The participant, in the opinion of the Investigator, is unable to adhere to the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (15):
- United States (9):
  - Orange, California
  - Gainesville, Florida
  - Kansas City, Kansas
  - St Louis, Missouri
  - New York, New York
  - Durham, North Carolina
  - Colombus, Ohio
  - Heshey, Pennsylvania
  - Fairfax, Virginia
- Germany (3):
  - Mainz
  - München
  - Münster
- Rotterdam, Netherlands
- United Kingdom (2):
  - Newcastle upon Tyne
  - Salford

REFERENCES:
- [Derived] van der Ploeg A, Carlier PG, Carlier RY, Kissel JT, Schoser B, Wenninger S, Pestronk A, Barohn RJ, Dimachkie MM, Goker-Alpan O, Mozaffar T, Pena LD, Simmons Z, Straub V, Guglieri M, Young P, Boentert M, Baudin PY, Wens S, Shafi R, Bjartmar C, Thurberg BL. Prospective exploratory muscle biopsy, imaging, and functional assessment in patients with late-onset Pompe disease treated with alglucosidase alfa: The EMBASSY Study. Mol Genet Metab. 2016 Sep;119(1-2):115-23. doi: 10.1016/j.ymgme.2016.05.013. Epub 2016 May 19. PMID 27473031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 centers between July 06, 2011 and December 19, 2013.
Period: Overall Study
Arm/Group | Alglucosidase Alfa
Started | 16
Full Analysis Set (FAS) | 16 (All participants who received at least 1 complete infusion of alglucosidase alfa.)
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: FAS population included all participants who received at least one complete infusion of alglucosidase alfa.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tissue Glycogen Content in Quadriceps Muscle Biopsy Samples at Week 26
Description: Tissue glycogen content was measured by quadriceps biopsies as 'percent area of tissue occupied by glycogen'.
Time Frame: Baseline, Week 26
Population: FAS population included all participants who received at least one complete infusion of alglucosidase alfa. Here, n = number of participants with both Baseline and Week 26 assessment of tissue glycogen content.
Measure: Mean (Standard Deviation); unit: percent area occupied by glycogen
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 16
percent area occupied by glycogen
  Baseline (n=14) | 5.3 (4.59)
  Change at Week 26 (n=13) | -1.6 (4.11)
Statistical Analysis 1: Comparison: Alglucosidase Alfa; Statistical significance for change from Baseline was measured using one sample t-test; Test type: Superiority or Other; p = 0.1860, one sample t-test

2. Secondary Outcome: Glycogen Distribution
Time Frame: Baseline, Week 26
Population: No quantitative data could be reported for this outcome as the assessment was qualitative in nature.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 0

3. Secondary Outcome: Muscle Fiber Morphology
Time Frame: Baseline, Week 26
Population: No quantitative data could be reported for this outcome as the assessment was qualitative in nature.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 0

4. Secondary Outcome: Lysosomal Inclusions
Time Frame: Baseline, Week 26
Population: No quantitative data could be reported for this outcome as the assessment was qualitative in nature.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 0

5. Secondary Outcome: Percent Change From Baseline in Muscle Involvement Using Mercuri Scoring at Week 26
Description: Muscle involvement was assessed by T1-weighted magnetic resonance imaging (MRI). T1-weighted MRI data was analyzed using the Mercuri scoring in both legs (Total score = 1-4; where 1=Normal appearance, 2=Mild involvement, 3=Moderate involvement, and 4=Severe involvement). For each participants, the average for each the upper (thigh) and lower leg was computed for Mercuri grading.
Time Frame: Baseline, Week 26
Population: FAS population included all participants who received at least one complete infusion of alglucosidase alfa. Here, Number of participants analyzed= participants with both Baseline and Week 26 assessment of muscle involvement, n= number of participants with both Baseline and Week 26 assessment of muscle involvement for specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 14
percent change
  Mercuri Scoring - Upper Leg (n=13) | 2.6 (9.24)
  Mercuri Scoring - Lower Leg (n=14) | 0.0 (0.0)

6. Secondary Outcome: Percent Change From Baseline in Degree of Fatty Infiltration Using 3-Point 3-Dimensional (3D) Dixon at Week 26
Description: Degree of Fatty Infiltration was assessed by 3-point 3D Dixon acquisition using skeletal muscle MRI in a subset of participants.
Time Frame: Baseline, Week 26
Population: FAS population included all participants who received at least one complete infusion of alglucosidase alfa. Here, number of participants analyzed = number of participants with both Baseline and Week 26 assessment of degree of fatty infiltration.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 3
percent change | 2.0 (12.83)

7. Secondary Outcome: Percent Change From Baseline in Disease Activity Using T2 Magnetic Resonance Imaging (MRI) at Week 26
Description: Disease activity (inflammation and/or water content within muscles) was quantitatively assessed by T2 MRI values in a subset of participants. A T2 MRI value of greater than (>) 39 millisecond (ms) was defined as abnormal. T2 estimation normally requires an additional acquisition for computing the B1 spatial deviation however, can still be estimated if this acquisition is missing.
Time Frame: Baseline, Week 26
Population: FAS population included all participants who received at least one complete infusion of alglucosidase alfa. Here Number of participants analyzed = number of participants with both baseline and Week 26 assessment of disease activity.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 6
percent change
  T2 with B1 | 8.1 (14.19)
  T2 without B1 | 7.2 (13.58)

ADVERSE EVENTS:
Time Frame: From signature of the informed consent form up to the final visit (Week 26)
Description: In the event a single participant has experienced both serious and non-serious form of the same adverse event (AE), individual has been included in numerator of both AE tables. Analysis was performed on the safety population: all participant who received any amount of alglucosidase alfa. AEs are listed independent of relationship to treatment.
Arm/Group | Alglucosidase Alfa
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=16)
Retinal vascular thrombosis (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=16)
Bradycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 1
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site extravasation (General disorders) | 1
Malaise (General disorders) | 1
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Heart rate increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Muscle contractions involuntary (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Epididymitis (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.